CLINICAL TRIAL: NCT00813982
Title: Daily Wear Comparison of Enhanced and Non-Enhanced Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-335-C-009
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Experimental Lotrafilcon A Contact Lens (Experimental): Lotrafilcon A experimental contact lens randomly assigned to one eye
  Interventions: Device: Lotrafilcon A Experimental Contact Lens
- Commercial Lotrafilcon A Contact Lens (Active Comparator): Lotrafilcon A commercial contact lens randomly assigned to one eye
  Interventions: Device: Lotrafilcon A Commercial Contact Lens

INTERVENTIONS:
Device: Lotrafilcon A Experimental Contact Lens — Experimental spherical, silicone hydrogel soft contact lens
  Arms: Experimental Lotrafilcon A Contact Lens
Device: Lotrafilcon A Commercial Contact Lens — Commercially marketed spherical, silicone hydrogel soft contact lens
  Arms: Commercial Lotrafilcon A Contact Lens

SUMMARY:
The purpose of this study is to compare an experimental contact lens with a currently marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Able to wear contact lenses for a minimum of 5 days a week, at least 8 hours a day
* On exam have ocular findings that are considered normal and would not prevent the safe wear of contact lenses
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* Requires concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Evidence of systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of their accessory solutions
* Any active corneal infection
* Any use of medications for which contact lens wear would be contraindicated
* History of corneal refractive surgery
* Wears toric contact lenses
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but not dispensed due to failing inclusion criteria. This participant is included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Groups:
- Experimental Contact Lens / Commercial Contact Lens: Lotrafilcon A experimental contact lens randomly assigned to one eye, with Lotrafilcon A commercial contact lens assigned to the fellow eye for contralateral wear.
Period: Overall Study
Arm/Group | Experimental Contact Lens / Commercial Contact Lens
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Contact Lens / Commercial Contact Lens
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: Overall vision was interpreted by the subject and recorded on a questionnaire as a single, retrospective evaluation of 1-week wear time. Overall vision was evaluated by eye and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week
Population: Per Protocol. Two participants were excluded from analysis due to major protocol deviations as determined by masked review. One participant was not analyzed due to discontinuation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Lotrafilcon A Commercial Contact Lens: Commercial spherical silicone hydrogel contact lens worn for one week on the same basis as habitual lenses -- ie., either on a daily wear or extended wear modality.
- Lotrafilcon A Experimental Contact Lens: Experimental spherical silicone hydrogel contact lens worn for one week on the same basis as habitual lenses -- ie., either on a daily wear or extended wear modality.
Arm/Group | Lotrafilcon A Commercial Contact Lens | Lotrafilcon A Experimental Contact Lens
Number analyzed (Participants) | 56 | 56
Units on a Scale | 8.7 (1.5) | 8.7 (1.7)

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Lotrafilcon A Commercial Contact Lens: Commercial spherical silicone hydrogel contact lens
- Lotrafilcon A Experimental Contact Lens: Experimental spherical silicone hydrogel contact lens
Arm/Group | Lotrafilcon A Commercial Contact Lens | Lotrafilcon A Experimental Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any pre-clinical and/or clinical data or impressions from this trial.